CLINICAL TRIAL: NCT03504488
Title: A Phase 1/2 Safety and Efficacy Dose Escalation / Dose Expansion Study of a CAB-ROR2-ADC, Alone and in Combination With a PD-1 Inhibitor, in Patients With Advanced Solid Tumors (Ph1) and Melanoma and NSCLC Patients (Ph2)
Brief Title: CAB-ROR2-ADC Safety and Efficacy Study in Patients With TNBC or Head & Neck Cancer (Ph1) and NSCLC or Melanoma (Ph2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA3021-001
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer; Triple Negative Breast Cancer; Melanoma; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Melanoma; Head and Neck Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy - CAB-ROR2-ADC (BA3021) alone (Experimental): BA3021 alone Q2W dosing regimen
  Interventions: Biological: CAB-ROR2-ADC
- Combination Therapy (Experimental): CAB-ROR2-ADC (BA3021) with PD-1 inhibitor
  Interventions: Biological: CAB-ROR2-ADC; Biological: PD-1 inhibitor

INTERVENTIONS:
Biological: CAB-ROR2-ADC — Conditionally active biologic anti-ROR2 antibody drug conjugate
  Other Names: BA3021
Biological: PD-1 inhibitor — PD-1 inhibitor
  Arms: Combination Therapy

SUMMARY:
The objective of this study is to assess safety and efficacy of CAB-ROR2-ADC in solid tumors

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase 1/2 study designed to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of BA3021, a conditionally active biologic (CAB) ROR2-targeted antibody drug conjugate (CAB-ROR2-ADC) BA3021 in patients with advanced solid tumors.

This study will consist of a dose escalation phase and a dose expansion phase with BA3021 in Phase 1. Phase 2 will study BA3021 alone or in combination with a PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumor and have failed all available standard of care (SoC) therapy and for whom no curative therapy is available or who are not eligible, intolerant to or refuse standard therapy.
* Patients must have measurable disease.
* For the dose expansion phase: Patients with locally advanced unresectable or metastatic, non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC) and soft tissue sarcoma (STS)
* Age ≥ 18 years.
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least three months.

Exclusion Criteria:

* Patients must not have clinically significant cardiac disease.
* Patients must not have known non-controlled CNS metastasis.
* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as wellas known or suspected allergy or intolerance to any agent given during this study.
* Patients must not have had major surgery within 4 weeks before first BA3021 administration.
* Patients must not have had prior therapy with a conjugated or unconjugated auristatin derivative/vinca-binding site targeting payload.
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety Profile | Up to 24 months
  Assess dose limiting toxicity as defined in the protocol
Phase 1: Safety Profile | Up to 24 months
  Assess maximum tolerated dose as defined in the protocol
Phase 1 and 2: Safety Profile | Up to 24 months
  Frequency and severity of AEs and/or SAEs
Phase 2: Confirmed Objective Response Rate (ORR) | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetics | Up to 24 months
  Plasma concentrations of ADC, total antibody and MMAE
Phase 1: Pharmacokinetics | Up to 24 months
  Peak Plasma Concentration (Cmax)
Phase 1: Pharmacokinetics | Up to 24 months
  Area under the plasma concentration versus time curve
Phase 1: Confirmed Objective Response Rate (ORR) | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR
Phase 1: Immunogenicity | Up to 24 months
  The number and percentage of patients who develop detectable anti-drug antibodies (ADAs)
Phase 1 and 2: Duration of response (DOR) | Up to 24 months
  Time from the first documented OR until the first documented disease progression or death (due to any cause), whichever occurs first
Phase 1 and 2: Progression-free survival (PFS) | Up to 24 months
  Time from the first dose of IP until the first documentation of disease progression or death due to any cause, whichever occurs first
Phase 1 and 2: Best overall response (OR) | Up to 24 months
  All post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy
Phase 1 and 2: Disease control rate (DCR) | Up to 24 months
  Proportion of patients with a best overall response of confirmed CR, confirmed PR, or stable disease (SD) ≥ 12 weeks
Phase 1 and 2: Time to response (TTR) | Up to 24 months
  Time from the first dose of investigational product until the first documentation of OR
Phase 1 and 2: Overall survival (OS) | Up to 24 months
  Time from the first dose of BA3021 treatment until death due to any cause
Phase 1 and 2: Tumor size | Up to 24 months
  Percent change from baseline in tumor size

CONTACTS AND LOCATIONS:
Locations (59):
- United States (38):
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope - Duarte, Duarte, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - California Research Institute, Los Angeles, California
  - USC Norris, Los Angeles, California
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Francisco, San Francisco, California
  - American Institute of Research, Whittier, California
  - University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute at Health One, Denver, Colorado
  - Florida Cancer Specialists & Research Institute, Fleming Island, Florida
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Memorial Cancer Institute (MCI), Hollywood, Florida
  - Florida Cancer Specialist - North, St. Petersburg, Florida
  - Memorial Sloan-Kettering Cancer Center, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Augusta University - Georgia Cancer Center, Augusta, Georgia
  - Baptist Health Systems, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Hematology/Oncology Clinic, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Care of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Roswell Park, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina- Hollings Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
- Greece (4):
  - HENRY DUNANT Hospital Center, 4th Department of Medical Oncology and Clinical Trials Unit, Athens
  - Metropolitan Hospital "Perseus Healthcare Group SA" 4th Oncology Department, Piraeus
  - Bioclinic Thessaloniki, Οncology Department, Thessaloniki
  - European Interbalkan Medical Center, Οncology Department, Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Poland (5):
  - MED-Polonia, Sp. z o.o. (LLC), Poznan, Greater Poland Voivodeship
  - Institute of Genetics and Immunology GENIM LCC in Lublin, Lublin, Lublin Voivodeship
  - Malgorzata Kozlik, Warsaw, Masovian Voivodeship
  - Polish Mother's Memorial Hospital-Research Institute, Lodz, Łódź Voivodeship
  - Beata Głogowska, Tomaszów Mazowiecki, Łódź Voivodeship
- Spain (6):
  - University Hospital Nuestra Senora de Valme, Seville, Andalusia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Anna Ramos Luna, Barcelona, Catalonia
  - University Clinic of Navarra - Madrid, Madrid
  - University Hospital 12 de Octubre, Madrid
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - LinKou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided